CLINICAL TRIAL: NCT01014273
Title: An International Randomized Trial of Trans-radial Versus Trans-femoral PCI Access Site Approach in Patients With Unstable Angina or Myocardial Infarction Managed With an Invasive Strategy. An Extension to the CURRENT (OASIS 7) Substudy (EFC5695): Effect of Type of Access for PCI (Radial or Femoral) on Bleeding Rate-Substudy.
Brief Title: A Trial of Trans-radial Versus Trans-femoral Percutaneous Coronary Intervention (PCI) Access Site Approach in Patients With Unstable Angina or Myocardial Infarction Managed With an Invasive Strategy
Acronym: RIVAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sanjit Jolly, MD, MSc, FRCPC, Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rad-Fem PCI Access Study
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-02

CONDITIONS: Acute Coronary Syndrome; Percutaneous Coronary Intervention
Keywords: Acute Coronary Syndrome; PCI; Percutaneous Coronary Intervention; Radial Access
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trans-femoral access (Active Comparator): Femoral artery PCI access site
  Interventions: Procedure: Percutaneous Coronary Intervention
- Trans-radial access (Active Comparator): Radial artery PCI access site
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention

SUMMARY:
This is a multi-national, multi-centre, randomized study comparing the trans-radial PCI access strategy and the trans-femoral PCI access strategy in ACS patients with UA or NSTEMI or STEMI planned to be treated with an invasive strategy (PCI).

The hypothesis is that radial access site PCI will be associated with significantly less major bleeding and access site complications compared with a femoral approach, without increasing the risk of ischemic events. The overall benefit-risk profile will favor a trans-radial approach.

ELIGIBILITY:
INCLUSION CRITERIA

1.1 UA/NSTEMI patients

Ischemic symptoms suspected to represent a non-ST segment elevation ACS (unstable angina [UA] or non-ST segment elevation myocardial infarction NSTEMI) defined as:

Clinical history consistent with new onset, or a worsening pattern, of characteristic ischemic chest pain occurring at rest or with minimal exercise (lasting longer than 10 minutes) and planned to be managed with an invasive strategy

AND at least one of the following:

1. Electrocardiogram (ECG) changes compatible with new ischemia [ST depression of at least 1mm or transient ST elevation or ST elevation of less than or equal to 1 mm or T wave inversion greater than 2 mm in at least 2 contiguous leads].

   or
2. Patients > 60 years of age with normal ECG are eligible provided there is a high degree of certainty that presenting symptoms are due to myocardial ischemia. Such patients must have documented evidence of previous coronary artery disease (CAD) with at least one of the following:

   * Prior MI requiring hospitalization
   * Prior revascularization procedure (more than 3 months ago)
   * Cardiac catheterization showing significant CAD
   * Positive exercise test
   * Other objective evidence of atherosclerotic vascular disease or
3. Already elevated cardiac enzymes or troponin I or T above the upper limit of normal.

1.2 STEMI patients

1. Presenting with signs or symptoms of acute myocardial infarction lasting at least 20 minutes and planned to be managed with an invasive strategy with intent to perform a percutaneous coronary intervention (PCI) during the index hospitalization.
2. Definite ECG changes compatible with STEMI: persistent ST-elevation (> 2 mm in two contiguous precordial leads or > 1 mm in at least two limb leads), or new left bundle branch block, or Q-wave in 2 contiguous leads

   2) Randomized during index hospitalization for acute coronary syndrome 3) Suitable candidate for either radial or femoral artery PCI 4) Intent to perform same-sitting angiography and PCI. 5) Palpable radial artery with documented normal Allen's test 6) Acceptance by operator to use whichever route is assigned by the randomization process 7) Previous experience of the operator with at least 50 cases of radial artery access within the past year 8) Written informed consent

   EXCLUSION CRITERIA
   1. Age < 18 years
   2. Active bleeding or significant increased risk of bleeding, severe hepatic insufficiency, current peptic ulceration, proliferative diabetic retinopathy.
   3. Uncontrolled hypertension
   4. Cardiogenic shock
   5. Prior CABG surgery with use of more than one internal mammary artery
   6. Documented severe peripheral vascular disease precluding a femoral approach
   7. Participation in any study with an investigational drug or device within the previous 30 days
   8. Medical, geographic or social factors making study participation impractical

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7021 (Actual)
Dates: Start 2006-06; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
First occurrence of the composite of death, MI, stroke or non CABG major bleeding (i.e. severe bleeding, other major bleeding) at 30 days. | 30 days

SECONDARY OUTCOMES:
Non CABG major bleeding | within 30 days following randomization
Death, MI or stroke | within 30 days following randomization

CONTACTS AND LOCATIONS:
Overall Officials: Sanjit Jolly, MD, MSc, FRCPC, Principal Investigator — Population Health Research Institute; Susan Chrolavicius, Study Director — Population Health Research Institute; Shamir Mehta, MD, MSc, FRCP(C), FACC, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Cantor WJ, Mehta SR, Yuan F, Dzavik V, Worthley M, Niemela K, Valentin V, Fung A, Cheema AN, Widimsky P, Natarajan M, Jedrzejowski B, Jolly SS. Radial versus femoral access for elderly patients with acute coronary syndrome undergoing coronary angiography and intervention: insights from the RIVAL trial. Am Heart J. 2015 Nov;170(5):880-6. doi: 10.1016/j.ahj.2015.08.011. Epub 2015 Aug 16. PMID 26542495
- [Derived] Jolly SS, Cairns J, Yusuf S, Niemela K, Steg PG, Worthley M, Ferrari E, Cantor WJ, Fung A, Valettas N, Rokoss M, Olivecrona GK, Widimsky P, Cheema AN, Gao P, Mehta SR; RIVAL Investigators. Procedural volume and outcomes with radial or femoral access for coronary angiography and intervention. J Am Coll Cardiol. 2014 Mar 18;63(10):954-63. doi: 10.1016/j.jacc.2013.10.052. Epub 2013 Nov 21. PMID 24269362
- [Derived] Jolly SS, Cairns J, Niemela K, Steg PG, Natarajan MK, Cheema AN, Rao SV, Cantor WJ, Dzavik V, Budaj A, Sheth T, Valentin V, Fung A, Widimsky P, Ferrari E, Gao P, Jedrzejowski B, Mehta SR; RIVAL Investigators. Effect of radial versus femoral access on radiation dose and the importance of procedural volume: a substudy of the multicenter randomized RIVAL trial. JACC Cardiovasc Interv. 2013 Mar;6(3):258-66. doi: 10.1016/j.jcin.2012.10.016. PMID 23517837
- [Derived] Mehta SR, Jolly SS, Cairns J, Niemela K, Rao SV, Cheema AN, Steg PG, Cantor WJ, Dzavik V, Budaj A, Rokoss M, Valentin V, Gao P, Yusuf S; RIVAL Investigators. Effects of radial versus femoral artery access in patients with acute coronary syndromes with or without ST-segment elevation. J Am Coll Cardiol. 2012 Dec 18;60(24):2490-9. doi: 10.1016/j.jacc.2012.07.050. Epub 2012 Oct 24. PMID 23103036
- [Derived] Jolly SS, Yusuf S, Cairns J, Niemela K, Xavier D, Widimsky P, Budaj A, Niemela M, Valentin V, Lewis BS, Avezum A, Steg PG, Rao SV, Gao P, Afzal R, Joyner CD, Chrolavicius S, Mehta SR; RIVAL trial group. Radial versus femoral access for coronary angiography and intervention in patients with acute coronary syndromes (RIVAL): a randomised, parallel group, multicentre trial. Lancet. 2011 Apr 23;377(9775):1409-20. doi: 10.1016/S0140-6736(11)60404-2. Epub 2011 Apr 4. PMID 21470671
- [Derived] Jolly SS, Niemela K, Xavier D, Widimsky P, Budaj A, Valentin V, Lewis BS, Avezum A, Steg PG, Rao SV, Cairns J, Chrolavicius S, Yusuf S, Mehta SR. Design and rationale of the radial versus femoral access for coronary intervention (RIVAL) trial: a randomized comparison of radial versus femoral access for coronary angiography or intervention in patients with acute coronary syndromes. Am Heart J. 2011 Feb;161(2):254-260.e1-4. doi: 10.1016/j.ahj.2010.11.021. PMID 21315206